CLINICAL TRIAL: NCT07401823
Title: An Open-Label Extension Study to Evaluate Long-Term Safety and Tolerability of Pociredir in Participants With Sickle Cell Disease (SCD) Who Have Participated in a Pociredir Study
Brief Title: Open-Label Extension Study to Pioneer Study 6058-SCD-101
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6058-SCD-102
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
Keywords: FTX-6058; Pociredir; Fetal hemoglobin; Sickle Cell Disease; Open-label; Anemia, Sickle Cell; Hematologic diseases
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pociredir (Experimental): Participants will receive Pociredir orally once daily (QD)
  Interventions: Drug: Pociredir

INTERVENTIONS:
Drug: Pociredir — Pociredir Oral Capsules will be administered
  Other Names: FTX-6058

SUMMARY:
This is an open-label study to evaluate the safety and tolerability of long-term treatment with pociredir without a comparator in participants with SCD who have previously been treated and shown benefit with pociredir in feeder study 6058-SCD-101 (NCT05169580). Participants in this study will receive once daily doses of pociredir for up to 48 months.

DETAILED DESCRIPTION:
The first dose of study drug will be administered on Day 1 in the clinic and participants will continue at home dosing once daily (QD). Dosing will occur in the clinic on days where there are clinic visits. Treatment Period clinic visits are planned every other week through Week 12 (Weeks 2, 4, 6, 8, 10, and 12), monthly through Week 24 (Weeks 16, 20, and 24), and then every 12 weeks from Week 24 through Week 192. A final follow-up visit (Week 196) will occur 4 weeks after the final dose of study drug at Week 192.

Participants will receive pociredir at the dose level they received in Study 6058-SCD-101 through Week 192, unless data from that study indicates a change to a different optimized dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 years and older must have previously participated in and successfully completed Study 6058-SCD-101.
* Participant has signed and dated the informed consent form (ICF) before any study-specific procedures are performed and is willing and able to comply with the study procedures and restrictions.
* Participants who meet all other inclusion and exclusion criteria for this study, and per Investigator's recommendation may continue standard of care as indicated with the exception of hydroxyurea (HU). Participants may continue crizanlizumab, and/or L-glutamine, but must be on a stable dose for at least 6 months.
* Participants, who if female and of childbearing potential, agree to use 2 effective methods of contraception, 1 of which must be highly effective, or practice abstinence starting at the time of the ICF signing to 90 days after the last dose of study drug, and, who if male, should use condoms or practice abstinence from the time of ICF signing to 90 days after the last dose of study drug.
* Documented HbF benefit, as judged by the Investigator, from prior study.
* Participant must meet both of the following laboratory values during Screening:

  1. Absolute neutrophil count ≥ 1.5 × 10^9/liter,
  2. Platelets ≥ 80 × 10^9/liter
* Absolute reticulocyte count during Screening > 100 × 10^9/liter.

Exclusion Criteria:

* Major surgery, serious illness (acute or chronic), infection (clinically significant bacterial, fungal, parasitic or viral infection which requires therapy), fever not resolved within 3 days of onset and requiring treatment, significant bleeding, cerebrovascular accident, or seizure within 14 days prior to signing the ICF and 14 days prior to starting study drug.
* Sickle cell complication requiring more than 24-hour care from a medical provider in hospital or emergency care setting in the 14 days prior to starting study drug.
* Use of medications that are moderate or strong inducers or inhibitors of cytochrome P450 (CYP) 3A4 or CYP2C8, inhibit P-glycoprotein, breast cancer resistance protein, or multidrug and toxin extrusion protein 2-K, or are substrates of CYP2B6 within 14 days prior to first dose of study drug or anticipated need for any of these medications during the study.
* Participation in any other study with an investigational agent other than pociredir within the past 60 days prior to the first dose of study drug.
* History of bone marrow transplant or hematopoietic stem cell transplant or gene therapies.
* Vaccination in the previous 7 days prior to the first dose of study drug.

Note: Other protocol specified criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-02-04 (Estimated); Study Completion 2030-07-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting Treatment Emergent Adverse Events (TEAEs) | Up to Week 196
Number of participants with clinically significant changes in 12-lead Electrocardiogram (ECGs) | Up to Week 196
Number of participants with clinically significant changes in Vital signs | Up to Week 196
Number of participants with clinically significant changes in Clinical laboratory tests | Up to Week 196
  Laboratory assessments including hematology, coagulation, serum chemistry and electrolytes, lipid panel, SCD characterization, serology, urinalysis and pregnancy tests will be performed.

SECONDARY OUTCOMES:
Change from Baseline in percent Fetal hemoglobin (HbF) | Baseline (Day 1), and Up to Week 192
Change from Baseline in percent Reticulocytes | Baseline (Day 1), and Up to Week 192
Change from Baseline in Red cell distribution width | Baseline (Day 1), and Up to Week 192
Change from Baseline in Unconjugated bilirubin | Baseline (Day 1), and Up to Week 192
Change from Baseline in Lactate dehydrogenase (LDH) | Baseline (Day 1), and Up to Week 192
Change from Baseline in Haptoglobin | Baseline (Day 1), and Up to Week 192
Change from Baseline in Reticulocyte count | Baseline (Day 1), and Up to Week 192
Number of participants reporting SCD-related complications | Up to Week 192
Annualized rate of Vaso-occlusive episode (VOE) | through end of month 48

IPD SHARING:
Plan to Share IPD: No